CLINICAL TRIAL: NCT01364961
Title: The Effects of Resveratrol on Serum Apolipoprotein A-I Concentrations in Men and Women With Low HDL-cholesterol Concentrations
Brief Title: Resveratrol and Serum Apo A-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: MEC 10-3-054
Record Dates: First submitted 2011-01-17; First posted 2011-06-03 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Dyslipidemia
Keywords: Resveratrol; FMD; PWV; HDL-cholesterol; Macrovasculature; Microvasculature
MeSH Terms: conditions — Dyslipidemias | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cellulose capsules (Placebo Comparator)
  Interventions: Dietary Supplement: Resveratrol capsules
- Resveratrol capsules (Experimental)
  Interventions: Dietary Supplement: Resveratrol capsules

INTERVENTIONS:
Dietary Supplement: Resveratrol capsules — 2 x 75 mg resveratrol each day, for 4 weeks
  Other Names: Resveratrol will be provided as resVida®

SUMMARY:
Although much effort has been done to lower LDL-cholesterol concentrations, there is still a substantial risk for cardiovascular disease (CVD). Another strategy to lower the risk for CVD is elevating the HDL-cholesterol (HDL-C). Both in vitro and in vivo studies showed that elevating HDL-C or apolipoprotein A-I (Apo A-I) levels protect against CVD. However, despite many initiatives, no new widely applicable intervention strategies with proven efficacy have been developed.

Epidemiologic studies have shown that a higher polyphenol intake is associated with a lower risk for CVD. Resveratrol, a polyphenol, could, through several beneficial mechanisms, exert a positive effect on formation of atherosclerotic plaques and thus on developing CVD. It has been shown in animals that resveratrol elevates PPAR-alpha activity. This may lead to elevated apo A-I and HDL-C levels in the blood. However, these effects are not shown in human intervention studies.

ELIGIBILITY:
Inclusion Criteria:

* aged between 45 and 70 years
* HDL-C <1.0 mmol/L (men)
* HDL-C <1.3 mmol/L (women)
* serum total cholesterol <8.0 mmol/L
* plasma glucose <7.0 mmol/L
* BMI between 25 - 35 kg/m2
* non-smoking
* willingness to abstain from resveratrol rich products from two weeks prior to the study and the duration of the study:

  * grapes and grape juice
  * wine (red and white)
  * all berries
  * peanuts
  * peanut butter
  * soy (products)
  * pomegranate

Exclusion Criteria:

* unstable body weight (weight gain or loss >3 kg in the past 3 months)
* indication for treatment with cholesterol-lowering drugs according to the Dutch Cholesterol Consensus
* use of medication or a medically-prescribed diet known to affect serum lipid or glucose metabolism
* Active cardiovascular disease (for instance congestive heart failure) or recent (<6 months) event, such as acute myocardial infarction or cerebro-vascular accident
* not willing to stop the consumption of vitamin supplements, fish oil capsules or products rich in plant stanol or sterol esters 3 weeks before the start of the study
* men: consumption of >21 glasses of alcohol-containing drinks per week women: consumption of >14 glasses of alcohol-containing drinks per week
* abuse of drugs
* pregnant or breastfeeding women
* participation in another biomedical study within 1 month prior to the screening visit
* having donated blood (as blood donor) within 1 month prior to the screening visit or planning to do so during the study
* impossible or difficult to puncture as evidenced during the screening visits

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
ApoA-I level | Measured at baseline, after 4 weeks, 8 weeks and 12 weeks

SECONDARY OUTCOMES:
Endothelial function and arterial stiffness | Measured in weeks 4 and 12
Endothelial function of the retinal microvasculature | Measured in weeks 4 and 12
Lipid and glucose metabolism during the fasting and postprandial phase | Measured at baseline, after 4 weeks, 8 weeks and 12 weeks
biomarkers for low-grade systemic inflammation and endothelial function | Measured at baseline, after 4 weeks, 8 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald P Mensink, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Derived] van der Made SM, Plat J, Mensink RP. Resveratrol does not influence metabolic risk markers related to cardiovascular health in overweight and slightly obese subjects: a randomized, placebo-controlled crossover trial. PLoS One. 2015 Mar 19;10(3):e0118393. doi: 10.1371/journal.pone.0118393. eCollection 2015. PMID 25790328